CLINICAL TRIAL: NCT06993142
Title: Slow-SPEED: Slowing Parkinson's Early Through Exercise Dosage
Acronym: Slow-SPEED
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: Stichting ParkinsonNL (Unknown); ZonMw: The Netherlands Organisation for Health Research and Development (Other); Michael J. Fox Foundation for Parkinson's Research (Other); Parkinson's UK (Other); Cure Parkinson's (Other); Edmond J. Safra Foundation (Unknown); Davis Phinney Foundation (Other); Sleep Medicine Centre Kempenhaeghe (Other); Sleep Medicine Centre SEIN (Unknown); Queen Mary University of London (Other); 23andMe, Inc. (Industry); Parkinsons Progression Markers Initiative (PPMI) (Unknown); Massachusetts General Hospital (Other); Harvard School of Public Health (HSPH) (Other); IJsfontein B.V., Netherlands (Unknown); Hoffmann-La Roche (Industry); Erasmus Medical Center (Other); University of Illinois at Chicago (Other); University of Rochester (Other); University of Bristol (Other); University of Plymouth (Other); University of Luebeck (Other); McGill University (Other); University of Pittsburgh (Other); Donders Centre for Cognitive Neuroimaging (Other); Parkinson's Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IRB ID: 13495; PF-Trail-1421986 (Other Grant/Funding Number: Parkinson's Foundation)
Record Dates: First submitted 2025-05-19; First posted 2025-05-28 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Parkinson Disease; Prodromal Stage; Neurodegenerative Diseases; Basal Ganglia Diseases; Central Nervous System Diseases; Synucleinopathies; Nervous System Diseases; Cerebral Disorder; Brain Diseases; Parkinsonian Disorders; Genetic Predisposition
Keywords: Physical activity; Prevention; Remote; Mobile Health (mHealth); Feasibility; Exercise; Digital biomarker; Motivational application; Walking; Parkinson Disease; Prodromal; LRRK2; GBA1; Genetic; Smartwatch
MeSH Terms: conditions — Parkinson Disease; Prodromal Symptoms; Neurodegenerative Diseases; Basal Ganglia Diseases; Central Nervous System Diseases; Synucleinopathies; Nervous System Diseases; Brain Diseases; Parkinsonian Disorders; Genetic Predisposition to Disease; Motor Activity

STUDY DESIGN:
Intervention Model Description: Parallel Assignment Double-blind randomized controlled trial
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Large increase in step count and moderate to vigorous physical activity relative to baseline level. (Experimental)
  Interventions: Behavioral: Increase of physical activity volume and intensity with the use of a motivational smartphone application
- Small increase in step count and moderate to vigorous physical activity relative to baseline level. (Active Comparator)
  Interventions: Behavioral: Increase of physical activity volume and intensity with the use of a motivational smartphone application

INTERVENTIONS:
Behavioral: Increase of physical activity volume and intensity with the use of a motivational smartphone application — A motivational smartphone application will be available for all participants using their own smartphone: the Slow-SPEED app. The Slow-SPEED app will motivate participants to increase the volume and intensity of their physical activity in daily life over a long period of time (2 years) based on their own baseline levels. Different treatment arms will receive different physical activity goals. The app offers participants feedback and support, that will stimulate them to reach their individual physical activity goal (i.e. incremental relative increase of step count and minutes exerting ≥ 64% of maximum heart rate reflecting moderate-to-vigorous physical activity (MVPA) relative to baseline level).

SUMMARY:
The goal of this clinical trial is two-fold. First to investigate the feasibility of whether a remotely administered smartphone app can increase the volume and intensity of physical activity in daily life in individuals with a LRRK2 G2019S or GBA1 N370S genetic mutation over a long period of time (24 months). Second, to explore the preliminary efficacy of exercise on markers for prodromal Parkinson's disease progression in individuals with a LRRK2 G2019S or GBA1 N370S genetic mutation.

Participants will be tasked to achieve an incremental increase of daily steps (volume) and amount of minutes exercised at a certain heart rate (intensity) with respect to their own baseline level. Motivation with regards to physical activity will entirely be communicated through the study specific Slow Speed smartphone app. A joint primary objective consists of two components. First to determine the longitudinal effect of an exercise intervention in LRRK2 G2019S or GBA1 N370S variant carriers on a prodromal load score, comprised of digital biomarkers of prodromal symptoms. The secondary component of the primary outcome is to determine the feasibility of a remote intervention study. The secondary objective is the effect of a physical activity intervention on digital markers of physical fitness. Exploratory outcomes entail retention rate, completeness of remote digital biomarker assessments, digital prodromal motor and non-motor features of PD. Using these biomarkers, the investigators aim to develop a composite score (prodromal load score) to estimate the total prodromal load. An international exercise study with fellow researchers in the United Kingdom are currently in preparation (Slow-SPEED-UK) and active in the Netherlands (Slow-SPEED-NL). Our intention is to analyse overlapping outcomes combined where possible through a meta-analysis plan, to obtain insight on (determinants of) heterogeneity in compliance and possible efficacy across subgroups

DETAILED DESCRIPTION:
Rationale: Parkinson's Disease (PD) is the fastest growing neurodegenerative disease. Exercise beneficially effects motor symptoms and neuroplasticity in people with PD. However, disease-slowing interventions have been ineffective in clinically manifest PD, when pathology is already advanced, but could succeed in prodromal PD, when pathology is limited. People with a LRRK2 G2019S or GBA1 N370S genetic mutation have an increased risk to develop clinically manifest PD. Therefore, this group is likely to develop prodromal PD. This study will take an important step forward by studying the feasibility and preliminary efficacy of long-term physical activity on prodromal symptoms and disease progression in people with prodromal PD using a newly developed, fully remote smartphone-based app. The app is inspired by the app used in the STEPWISE trial (NCT04848077) and currently used in Slow-SPEED-NL (NCT06193252).

Objective: The joint primary objective has two components. First, to evaluate the long-term (36-month) impact of an exercise intervention on a prodromal load score in individuals carrying the LRRK2 G2019S or GBA1 N370S variants. This score will be derived from digital biomarkers capturing both motor and non-motor prodromal symptoms. Using these biomarkers, the investigators aim to develop a composite prodromal load score to estimate the overall burden of prodromal features.

The secondary component of the primary outcome is to determine the feasibility of a long-term (36 months) remote intervention study expressed as longitudinal change in digital measures of physical activity (step count) measured using a Fitbit smartwatch.

Our secondary objective is the potential group effect on physical fitness. Thirdly, the investigators investigate whether the intervention, prodromal motor- and non-motor symptoms can be assessed remotely in a digital, decentralized fashion.

Currently blood- and imaging biomarkers are not incorporated as outcome measures. The investigators intend to add these biomarkers pending appropriate funding.

Study design: Double-blind randomized controlled trial

Study population: A total of 600 English speaking individuals living in the United States of America with a LRRK2 G2019S or GBA1 N370S genetic mutation aged 50 years and older, who are in possession of a suitable smartphone without mobility hampering conditions and absence of cognitive impairment which impedes usage of a smartphone will be recruited. Participant recruitment will primarily target individuals from the 23andMe customer base. Enrollment and onboarding of study participants will be supported by research staff at the University of Rochester.

Intervention: Participants will be randomized to a group (1:1 ratio) and will be motivated to increase the volume and intensity of physical activity based on their own baseline level. Baseline physical activity levels will be determined during a 4-week period. The two groups differ in the amount of physical activity that they are tasked to achieve.

ELIGIBILITY:
Inclusion criteria

1. previously identified LRRK2 G2019S or GBA N370S variant based on genotyping
2. aged 50 years or older
3. able to understand the English language
4. being able to walk independently inside the home without the use of a walking aid
5. in possession of a suitable smartphone (screen size minimum 4.6 inch), (Android version 9 or iOS version 15 or newer)
6. Not in a high physical activity range during the 4-week eligibility and baseline period

Exclusion criteria

1. clinically diagnosed or self-reported diagnosis neurodegenerative disease
2. self-reported falls of three or more per year
3. dexterity problems or cognitive impairments hampering smartphone use
4. if they are not aware of and do not wish to be informed about an increased risk of developing diseases associated with the LRRK2 or GBA1 risk variant
5. if individual is not community-dwelling
6. in possession of one of the following devices: Huawei P8 Lite; Huawei P9 Lite; Xiaomi Mi 6; Huawei P20 Lite (Fitbit is incompatible)

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2029-06-30 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in composite prodromal load score | From inclusion (week 0) to the end of treatment (week 156)
  Change in prodromal load score, comprised of digital biomarkers for prodromal symptoms. The score is currently under development.
Mean change in step count per day | All 4 week periods between and including week -4 until 0 (baseline period) and week 152 until 156 (end of treatment)
  Mean change in step count per day as measured continuously with a smartwatch. Mean steps per day will be calculated from 4-week periods. Higher positive change in step count indicate more volume of physical activity.

SECONDARY OUTCOMES:
Change in moderate to vigorous physical activity (MVPA) per day | All 4 week periods between and including week -4 until 0 (baseline period) and week 152 until 156 (end of treatment)
  Change in number of minutes exerting (minimally) ≥ 64% of maximum heart rate, reflecting moderate intense physical activity, measured continuously using a smartwatch. Mean minutes per day will be calculated from 4-week periods. Higher positive change in minutes of MVPA indicate more aerobic physical activity.
Change in resting heart rate (physical fitness) | All 4 week periods between and including week -4 until 0 (baseline period) and week 152 until 156 (end of treatment)
  Change in resting heart rate per day as measured continuously with a smartwatch. Mean resting heart rate per day will be calculated from 4-week periods. Higher negative change (i.e. lower resting heart rate) indicate better function.
Change in heart rate variability (physical fitness & autonomic function) | All 4 week periods between and including week -4 until 0 (baseline period) and week 152 until 156 (end of treatment)
  Change in heart rate variability in Root Mean Square of Successive Differences (RMSSD) measured every 5 minutes with a smartwatch. Mean RMSSD per day will be calculated from 4-week periods. Higher positive change in RMSSD indicate better function.
Change in VO2max (physical fitness) | All 4 week periods between and including week -4 until 0 (baseline period) and week 152 until 156 (end of treatment)
  Change in VO2max in ml/kg/min measured per day with a smartwatch. Mean VO2max per day will be calculated from 4-week periods. Higher positive change in VO2max indicate better function.
Change in anxiety and depression (HADS) | Week 0 (baseline), week 52 (1 year), week 104 (2 years), week 156 (end of treatment)
  Change from baseline (week 0) on the Hospital Anxiety and Depression Scale (HADS) at week 52 (1 year) and week 104 (2 years), and week 156 (end of treatment). Total range 0-42. Divided Anxiety and Depression scale have a range of 0-21. Higher scores indicate worse function.
Change in cognition (CANTAB web-version) | Week 0 (baseline), week 52 (1 year), week 104 (2 years), week 156 (end of treatment)
  Change from baseline (week 0) on the Cambridge Neuropsychological Test Automated Battery (CANTAB) at week 52 (1 year), week 104 (2 years) and week 156 (end of treatment). More errors indicate worse function.
Mean change in light sleep (sleep stage) | All 4 week periods between and including week -4 until 0 (baseline period) and week 152 until 156 (end of treatment)
  Mean change in light sleep stage measured continuously with a smartwatch. Mean duration of light sleep per day will be calculated from 4-week periods. Higher positive change indicate more light sleep.
Mean change in deep sleep (sleep stage) | All 4 week periods between and including week -4 until 0 (baseline period) and week 152 until 156 (end of treatment)
  Mean change in deep sleep stage measured continuously with a smartwatch. Mean duration of deep sleep per day will be calculated from 4-week periods. Higher positive change indicate more deep sleep.
Mean change in REM sleep (sleep stage) | All 4 week periods between and including week -4 until 0 (baseline period) and week 152 until 156 (end of treatment)
  Mean change in rapid eye movement (REM) sleep stage measured continuously with a smartwatch. Mean duration of REM sleep per day will be calculated from 4-week periods. Higher positive change indicate more REM sleep.
Change in self-reported sleep quality (PSQI) | Week 0 (baseline), week 52 (1 year), week 104 (2 years), week 156 (end of treatment)
  Change from baseline (week 0) on the Pittsburgh Sleep Quality Index (PSQI) at week 52 (1 year) and week 104 (2 years), and week 156 (end of treatment). Range 0-21. Higher scores indicate worse sleep quality.
Change in REM-sleep behavior disorder (RBDSQ) | Week 0 (baseline), week 52 (1 year), week 104 (2 years), week 156 (end of treatment)
  Change in question of the REM-sleep behavior disorder (RBD) single screening questionnaire (RBDSQ) at week 52 (1 year) and week 104 (2 years), and week 156 (end of treatment). 'Yes' indicates a higher likelihood of having RBD.
Change in olfaction (UPSIT) | Week 0 (baseline), week 156 (end of treatment)
  Change from baseline (week 0) on the University of Pennsylvania Smell Identification Test (UPSIT) at week 156 (end of treatment). Range 0-40. Higher scores indicate better function.
Change in motor symptoms (Roche PD Research mobile application) | Week 0, Week 6, Week 12, Week 18, Week 24, Week 30, Week 36, Week 42, Week 48, Week 54, Week 60, Week 66, Week 72, Week 78, Week 84, Week 90, Week 96, Week 102, Week 108, Week 114, Week 120, Week 126, Week 132, Week 138, Week 144, Week 150, Week 156
  Change in motor symptoms measured digitally with the smartphone using the Roche PD Research mobile application. Higher scores indicate worse function. 6-weekly testing interval. Optional to complete the tests weekly.
Change in instrumental activities of daily living (ADL) (functional status) | Week 0 (baseline), week 52 (1 year), week 104 (2 years), week 156 (end of treatment)
  Change from baseline (week 0) on Lawton instrumental ADL (iADL) scale at week 52 (1 year) and week 104 (2 years), and week 156 (end of treatment). Range 0-14. Higher score indicate better function.
Change in WHOQoL-BREF (quality of life) | Week 0 (baseline), week 52 (1 year), week 104 (2 years), week 156 (end of treatment)
  Change from baseline (week 0) on World Health Organization Quality of Life Questionnaire - BREF (WHOQoL-BREF) scale at week 52 (1 year) and week 104 (2 years), and week 156 (end of treatment). Range 0-100. Higher score indicate better quality of life.
Change in Research and Development (RAND-36)/Short Form health survey (SF-36) (quality of life) | Week 0 (baseline), week 52 (1 year), week 104 (2 years), week 156 (end of treatment)
  Change from baseline (week 0) on RAND-36/SF-36 scale at week 52 (1 year) and week 104 (2 years), and week 156 (end of treatment). Range 0-100. Higher score indicate better quality of life.
Change in MDS-UPDRS part 1b (Non-Motor Experiences of Daily Living) | Week 0 (baseline), week 52 (1 year), week 104 (2 years), week 156 (end of treatment)
  Change from baseline (week 0) on MDS-UPDRS part 1b scale at week 52 (1 year) and week 104 (2 years), and week 156 (end of treatment). Range 0-24. Higher score indicate worse function.
Change in MDS-UPDRS part 2 (Motor Experiences of Daily Living) | Week 0 (baseline), week 52 (1 year), week 104 (2 years), week 156 (end of treatment)
  Change from baseline (week 0) on MDS-UPDRS part 2 at week 52 (1 year) and week 104 (2 years), and week 156 (end of treatment). Range 0-56. Higher score indicate worse function.
System Usability (SUS) | Week 0 (baseline), week 52 (1 year), week 104 (2 years), week 156 (end of treatment)
  Usability of the Slow-SPEED smartphone application assessed by the System Usability Scale (SUS) at week 52 (1 year) and week 104 (2 years), and week 156 (end of treatment). Range 0-100. Higher score indicate better usability.
Barriers and motivators to engage in physical activity | Week 0 (baseline) and week 156 (end of treatment)
  Barriers and motivators to engage in physical activity reported on a self-developed questionnaire. Section 1: Exercise history (qualitative), section 2: Overall motivation to exercise (0-10, higher score indicates higher motivation), section 3: Specific motivations to exercise (0-14, higher score indicaties more motivational factors), Section 4: barriers to exercise (0-20, higher score indicates more barriers), Section 5: Main motivations and barriers to exercise (qualitative).
Change in phenoconversion neurodegenerative disease (0-100%) | Week 0 (baseline) and week 156 (end of treatment)
  Change from baseline (week 0) on phenoconversion in Parkinson's Disease (PD), Lewy body dementia (LBD) and multiple system atrophy (MSA) at week 156 (end of treatment). Higher scores indicate more phenoconversion.
Change in REM-sleep behavior disorder diagnosis | Week 0 (baseline) and week 156 (end of treatment)
  Change from baseline (week 0) on diagnoses of REM-sleep behavior disorder (rBD). Higher scores indicate more RBD diagnoses.
Change in step count on a group level (compliance) | Week -4 until 0 (baseline) compared to week 0-26, week 26-52, week 52-78, week 78-104, Week 104-130, Week 130-156
  Change from week -4 until 0 (baseline period) mean step count per day compared to mean step count in 6 month periods. Mean step count per day will be calculated from 4-week periods. Scored as number of participants able to increase step count per day 0-25%, 26-50%, 51-75%, 76-100% relative to their own baseline measure
Change in moderate to vigorous physical activity per day on a group level (compliance) | Week 0-26, Week 26-52, Week 52-78, Week 78-104, Week 104-130, Week 130-156
  Change from week -4 until 0 (baseline period) number of minutes exerting (minimally) ≥ 64% of maximum heart rate in 6 month periods. Mean minutes per day will be calculated from 4-week periods. Scored as number of participants to increase 0-25%, 26-50%, 51-75%, 76-100% relative to their own baseline measure
Number of completed step week goals on a group level (compliance) | Week 0 (baseline) and week 156 (end of treatment)
  Total number of completed step count week goals
Number of completed aerobic activity (MVPA intensity) week goals on a group level (compliance) | Week 0 (baseline) and week 156 (end of treatment)
  Total number of completed aerobic activity (MVPA intensity) week goals
Number of drop-outs on a group level (retention rate) | Week 0 (baseline), week 26, week 52, week 78, week 104, week 130, week 156 (end of treatment)
  Number of drop-outs throughout the study
Number of interactions with Slow-SPEED app on a group level | Week 0 (baseline), week 26, week 52, week 78, week 104, week 130, week 156 (end of treatment)
  Total times opening the app
Number of completed questionnaires on group level (completeness of digital assessments) | Week 0 (baseline), week 52 (1 year), week 104 (2 years), week 156 (end of treatment)
  Number of completed questionnaires
Number of smartwatch data points on group level (completeness of digital assessments) | Week 0 (baseline), week 26, week 52, week 78, week 104, week 130, week 156 (end of treatment)
  Number of data points received for each selected smartwatch parameter
Total smartwatch wear time on group level (completeness of digital assessments) | Week 0 (baseline), week 26, week 52, week 78, week 104, week 130, week 156 (end of treatment)
  Total smartwatch wear time
Number of Roche PD Research mobile application data points on group level (completeness of digital assessments) | Week 0, Week 6, Week 12, Week 18, Week 24, Week 30, Week 36, Week 42, Week 48, Week 54, Week 60, Week 66, Week 72, Week 78, Week 84, Week 90, Week 96, Week 102, Week 108, Week 114, Week 120, Week 126, Week 132, Week 138, Week 144, Week 150, Week 156
  Number of data points received

CONTACTS AND LOCATIONS:
Overall Officials: Sirwan KL Darweesh, PhD, Principal Investigator — Radboudumc Department of Neurology
Locations (2):
- University of Rochester Center for Health and Technology (CHeT), Rochester, New York, United States
- Radboud University Medical Center, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
We will make relevant anonymised data available in a database.
Supporting Information: Study Protocol
Time Frame: We will make relevant anonymised data available in a database after publication of the main results of our trial.
Access Criteria: Researchers who are interested in re-use of the data are asked to contact the central contact person for permission.